CLINICAL TRIAL: NCT02271230
Title: Intervention With Vitamin D and Omega-3 Supplements and Incident Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Luc Djousse, Director of Research, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014P001206
Record Dates: First submitted 2014-10-07; First posted 2014-10-22 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Vitamin D; Fish Oils; Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Vitamin D and fish oil (Experimental): 2000 IU per day and 1 g per day of fish oil
  Interventions: Drug: Vitamin D and fish oil
- Vitamin D alone (Placebo Comparator): 2000 IU Vitamin D and fish oil placebo
  Interventions: Drug: Vitamin D alone
- Fish oil (EPA/DHA) alone (Experimental): 1 g per day of fish oil and vitamin D placebo
  Interventions: Dietary Supplement: Fish oil (EPA/DHA) alone
- Fish oil and vitamin D placebo (Placebo Comparator): Placebo for both vitamin D and fish oil
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D and fish oil — 2000 IU vitamin D and 1g/d fish oil
  Arms: Vitamin D and fish oil
Dietary Supplement: Fish oil (EPA/DHA) alone — 1 g/d fish oil
  Arms: Fish oil (EPA/DHA) alone
Drug: Vitamin D alone — 2000 IU vitamin D
  Arms: Vitamin D alone
Other: Placebo — Vitamin D placebo and fish oil placebo
  Arms: Fish oil and vitamin D placebo

SUMMARY:
This study will examine whether an intervention with vitamin D or fish oil supplements can reduce the risk of heart failure among adult men and women during a follow up period of up to five years (starting from the time of randomization into the parent VITAL trial). The investigators hypotheses are that both vitamin D and fish oil supplements will each reduce the risk of heart failure.

DETAILED DESCRIPTION:
For this ancillary study of the ongoing parent VITAL trial, we will adjudicate incident heart failure cases occurring during a time period of up to five years starting from randomization of subjects in the parent VITAL study. Intention-to-treat analysis will be used to assess the efficacy of vitamin D as well as omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 50 or older or women aged 55 or older
* Be consuming no more than 800 IU of vitamin D from all supplemental sources combined (individual vitamin D supplements, calcium+vitamin D supplements, medications with vitamin D [e.g., Fosamax Plus D], and multivitamins), or, if taking, willing to decrease or forego such use during the trial;
* Be consuming no more than 1200 mg/d of calcium from all supplemental sources combined, or, if taking, willing to decrease or forego such use during the trial;
* Not be taking fish oil supplements, or, if taking, willing to forego their use during the trial

Exclusion Criteria:

* prevalent heart failure
* History of cancer (except non-melanoma skin cancer), heart attack, stroke, transient ischemic attack, angina pectoris, CABG, or PCI
* History of renal failure or dialysis, hypercalcemia, hypo- or hyperparathyroidism, severe liver disease (cirrhosis), or sarcoidosis or other granulomatous diseases such as active chronic tuberculosis or Wegener's granulomatosis;
* Allergy to fish or soy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2014-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 401605 adults were initially screened; 39430 eligible to enter run-in; 25871 eligible for randomization; 2x2 factorial design: 12927 assigned to active vit D (of these, 6463 were assigned to active omega-3 FAs and 6464 to placebo omega-3 FAs) & 12944 assigned to placebo vit D (of these, 6470 were assigned to active omega-3 FAs and 6474 to placebo omega-3 FAs)
Pre-assignment Details: The trial included a 3-month placebo run-in period to select participants likely to have excellent compliance. Only individuals who reported taking at least 2/3 of their study pills during the run-in and met other eligibility criteria were randomized into the trial.
Groups:
- Active Vitamin D + Active Omega-3 Fatty Acids: Active Vitamin D = Vitamin D3, one 2000 IU capsule/day; Active Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- Active Vitamin D + Placebo Omega-3 Fatty Acids: Active Vitamin D = Vitamin D3, one 2000 IU capsule/day; Placebo Omega-3 Fatty Acids, one capsule/day
- Placebo Vitamin D + Active Omega-3 Fatty Acids: Placebo Vitamin D, one capsule/day; Active Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- Placebo Vitamin D + Placebo Omega-3 Fatty Acids: Placebo Vitamin D, one capsule/day; Placebo Omega-3 Fatty Acids, one capsule/day
Period: Overall Study
Arm/Group | Active Vitamin D + Active Omega-3 Fatty Acids | Active Vitamin D + Placebo Omega-3 Fatty Acids | Placebo Vitamin D + Active Omega-3 Fatty Acids | Placebo Vitamin D + Placebo Omega-3 Fatty Acids
Started | 6463 | 6464 | 6470 | 6474
Completed | 6463 | 6464 | 6470 | 6474
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of participants enrolled in the VITAL-Heart Failure ancillary study stratified by randomization arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Vitamin D + Active Omega-3 Fatty Acids | Active Vitamin D + Placebo Omega-3 Fatty Acids | Placebo Vitamin D + Active Omega-3 Fatty Acids | Placebo Vitamin D + Placebo Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 6463 | 6464 | 6470 | 6474 | 25871
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.1) | 67.1 (7.0) | 67.2 (7.1) | 67.1 (7.1) | 67.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3276 | 3271 | 3271 | 3267 | 13085
  Male | 3187 | 3193 | 3199 | 3207 | 12786
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not all participants reported race/ethnicity Population: Not all participants provided information on race/ethnicity; hence the discrepancy between number reported under race/ethnicity and total number enrolled.
  Participants
    count: number analyzed (Participants) | 6329 | 6318 | 6324 | 6333 | 25304
    count: Non-Hispanic White | 4515 | 4498 | 4529 | 4504 | 18046
    count: African American | 1278 | 1275 | 1271 | 1282 | 5106
    count: Hispanic (not African American) | 246 | 270 | 245 | 252 | 1013
    count: Asian/Pacific Islander | 102 | 86 | 98 | 102 | 388
    count: Native American/Alaskan Native | 62 | 56 | 58 | 52 | 228
    count: Other/Unknown | 126 | 133 | 123 | 141 | 523
Region of Enrollment [Number; unit: participants]
  United States | 6463 | 6464 | 6470 | 6474 | 25871

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Heart Failure Hospitalization
Description: We will consider any hospitalization for heart failure among participants enrolled in the parent VITAL trial for this ancillary study. Incident heart failure are initially captured through annual questionnaires with subsequent validation by a team of physicians with expertise in cardiovascular medicine and epidemiology. We excluded 36 participants with prevalent heart failure at the time of randomization for the primary analysis.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin D: Vitamin D3, one 2000 IU capsule/day
- Vitamin D Placebo: Vitamin D placebo, one capsule/day
- Active Omega-3 Fatty Acids: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Omega-3 Fatty Acids Placebo: Omega-3 fatty acids placebo, one capsule/day
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12904 | 12931 | 12912 | 12923
Participants | 240 | 259 | 244 | 255
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.78 to 1.11]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.80 to 1.14]

2. Secondary Outcome: Number of Recurrent Heart Failure Hospitalization
Description: Recurrent heart failure hospitalizations ascertained either by review of medical records and/or use of CMS (Center for Medicare and Medicaid Services) data.
Time Frame: 5 years
Population: Each participant is allowed to have multiple heart failure hospitalizations.
Measure: Number; unit: hospitalizations for heart failure
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
hospitalizations for heart failure | 341 | 364 | 326 | 379
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.81 to 1.09]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 0.998]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Conditions monitored for Vit D: kidney stones, hypercalcemia, parathyroid disease, kidney failure or dialysis; Other symptoms/side effects: gastrointestinal (GI) bleed, easy bruising; stomach upset or pain; nausea; constipation, diarrhea, skin rash Conditions monitored for omega-3: GI bleed; blood in urine; easy bruising; nosebleeds; kidney failure or dialysis; Other side effects: stomach upset or pain; nausea; constipation; diarrhea; skin rash; bad taste in mouth; increased burping
Groups:
- Active Vitamin D: Vitamin D3, one capsule of 2,000 IU/day
- Vitamin D Placebo: Vitamin D placebo, 1 capsule/day
- Active Omega-3 Fatty Acids: Omacor, 1 g capsule/day Each capsule of Omacor contains 465 mg of eicosapentaenoic acid (EPA) and 375 mg of docosahexaenoic acid (DHA)
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
All-Cause Mortality (participants affected / at risk) | 485/12927 | 493/12944 | 493/12933 | 485/12938
Serious Adverse Events (participants affected / at risk) | 1673/12927 | 1659/12944 | 1613/12933 | 1619/12938
Other Adverse Events (participants affected / at risk) | 10086/12927 | 10098/12944 | 10094/12933 | 10090/12938
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D (N=12927) | Vitamin D Placebo (N=12944) | Active Omega-3 Fatty Acids (N=12933) | Omega-3 Fatty Acids Placebo (N=12938)
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 341 | 403 | 370 | 374
Hypercalcemia (Endocrine disorders) | 147 | 143 | 151 | 139
Invasive cancer of any type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 793 | 824 | 820 | 797
Death from cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 154 | 187 | 168 | 173
Breast cancer in women (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 124 | 122 | 117 | 129
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 192 | 219 | 219 | 192
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 | 47 | 54 | 44
Major cardiovascular events (Vascular disorders) | 396 | 409 | 386 | 419 — Composite of myocardial infarction, stroke, and cardiovascular death
Myocardial infarction (Vascular disorders) | 169 | 176 | 145 | 200
Stroke (Vascular disorders) | 141 | 149 | 148 | 142
Death from cardiovascular causes (Vascular disorders) | 152 | 138 | 142 | 148
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D (N=12927) | Vitamin D Placebo (N=12944) | Active Omega-3 Fatty Acids (N=12933) | Omega-3 Fatty Acids Placebo (N=12938)
Easy bruising (Blood and lymphatic system disorders) | 3434 | 3408 | 3443 | 3399
Frequent nosebleeds (Blood and lymphatic system disorders) | 466 | 490 | 465 | 491
Blood in urine (Blood and lymphatic system disorders) | 911 | 882 | 919 | 874
Parathyroid condition (Endocrine disorders) | 50 | 62 | 52 | 60 — hyperparathyroidism or hypoparathyroidism
Stomach upset or pain (Gastrointestinal disorders) | 4860 | 4870 | 4887 | 4843
Nausea (Gastrointestinal disorders) | 3519 | 3589 | 3558 | 3550
Constipation (Gastrointestinal disorders) | 5133 | 5162 | 5184 | 5111
Diarrhea (Gastrointestinal disorders) | 5511 | 5668 | 5599 | 5580
Increased burping (Gastrointestinal disorders) | 2168 | 2207 | 2217 | 2158
Bad taste in mouth (General disorders) | 2195 | 2290 | 2240 | 2245
Kidney stones (Renal and urinary disorders) | 477 | 426 | 430 | 473
Kidney failure or dialysis (Renal and urinary disorders) | 85 | 88 | 85 | 88
Skin rash (Skin and subcutaneous tissue disorders) | 3268 | 3430 | 3331 | 3367

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT02271230/Prot_SAP_000.pdf